CLINICAL TRIAL: NCT04106609
Title: Randomized, Controlled Trial of an Individualized Exercise Oncology Program for Newly Diagnosed Breast Cancer Patients
Brief Title: Individualized Exercise Oncology Program for Newly Diagnosed Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Wonders (Other)
Responsible Party: Sponsor-Investigator, Karen Wonders, Executive Director, Maple Tree Cancer Alliance, Kettering Health Network
Organization: Kettering Health Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Maple Tree Exercise
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Patients will complete a 60-minute exercise session once per week for 12 weeks. The exercise sessions will be individualized to the patient's needs and fitness level by a trainer. A patient will work with the same trainer throughout the study, who will plan the patient's individualized exercise regimen, and who will provide one-on-one supervision for the duration of each 60-minute session. Each 60-minute session will include cardiovascular, strength, and flexibility training. The intensity level for the aerobic exercise ranges from 30-45% of the individual's predicted VO2max, controlled by heart monitors and lasting 30 min. Strength training will involve a full body workout, with emphasis on all major muscle groups and employing machines, free weights, and resistance tubing. Patients will complete 3 sets of 10 repetitions for each strength exercise. Flexibility training will involve static stretching of all major muscle groups for 15-20 seconds at the completion of each workout.
  Interventions: Other: Supervised, individualized exercise oncology program
- Control Group (Active Comparator): The control group will receive the current standard of care, which includes a resource guide with various options available to the cancer survivor. Within this guide are tips for healthy eating and pictures of standard exercises to improve fitness.
  Interventions: Other: Current standard of care

INTERVENTIONS:
Other: Supervised, individualized exercise oncology program — The study intervention is a supervised, individualized exercise oncology program described in previous literature2,3,12 and provided by Maple Tree Cancer Alliance, a non-profit organization providing exercise training to individuals with cancer (https://www.mapletreecanceralliance.org/). This organization was founded in 2011 and currently operates in 9 hospitals serving Ohio and Pennsylvania, offering free exercise programs and nutritional guidance to approximately 500 patients annually to help relieve side effects related to cancer treatment.
  Arms: Exercise Group
Other: Current standard of care — Resource guide with various options available to cancer survivor. Within this guide are tips for healthy eating and pictures of standard exercises to improve fitness.
  Arms: Control Group

SUMMARY:
To test the effect of an individualized exercise oncology program on healthcare utilization, 30-day hospital readmission, pain, and cancer treatment tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Female; determined from electronic medical record
* Initial stage 0, 1 or 2 breast cancer diagnosis within the past 12 weeks determined from electronic medical record
* Age 30-80; determined from electronic medical record
* Physician clearance to participate in exercise

Exclusion Criteria:

* Participation in supervised physical exercise within 6 months prior to study enrollment
* Currently pregnant or planning to become pregnant
* Non-English speaking
* Unable to make own medical decisions and/or to follow verbal instructions

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Wonders, PhD, FACSM, Principal Investigator — Maple Tree Cancer Alliance
Locations (1):
- Maple Tree Cancer Alliance, Dayton, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Group: Supervised, individualized exercise oncology program: Patients in the supervised exercise intervention group completed 12 weeks of prescribed, individualized exercise that aligned with ACSM exercise guidelines for cancer survivors. Total dose of exercise was one time weekly, with cardiovascular, resistance training, and flexibility components. Cardiovascular exercise was performed on a treadmill. The intensity level for the aerobic exercise began with 30 min at 30% of the individual's predicted VO2max, assessed by heart monitors. Each week, intensity was progressed until the participant reached 45%. Strength training involved a full body workout, with emphasis on all major muscle groups and employed machines, free weights, and tubing. Patients completed 3 sets of 10 repetitions for each exercise. Each exercise program was individualized for each patient, but included the following resistance exercises: chest press, seated row, overhead press, leg extension, leg curl, leg press. Resistance intensity was set at a minimum of 30% of the individual's 1RM, or when the patient felt sufficiently fatigued after 10 repetitions completed with proper form. As the patient's RPE values decreased with each exercise, intensity was progressively increased, accordingly. Flexibility training involved static stretching of all major muscle groups for 15-20 seconds at the completion of each workout. Each session lasted approximately 60 minutes.
Period: Overall Study
Arm/Group | Exercise Group | Control Group
Started | 129 | 122
Completed | 123 | 120
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Group | Control Group | Total
Number analyzed (Participants) | 129 | 122 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (0.19) | 57.1 (0.15) | 56.45 (0.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 122 | 251
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 25
  Not Hispanic or Latino | 108 | 108 | 216
  Unknown or Not Reported | 7 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 9 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 21 | 38
  White | 80 | 78 | 158
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 14 | 35
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.74 (0.68) | 30.24 (0.56) | 29.48 (0.62)
Time Since Diagnosis [Mean (Standard Deviation); unit: months] | 1.2 (0.88) | 2.1 (0.82) | 1.65 (0.85)
Stage I Breast Cancer [Number; unit: participants] | 53 | 51 | 104
Stage II Breast Cancer [Number; unit: participants] | 76 | 71 | 147

OUTCOME MEASURES:

1. Primary Outcome: Missed Fractions
Description: Total number of missed fractions, determined by electronic medical record
Time Frame: 12 weeks
Population: This data was not collected from the medical record. Study personnel could not determine this from the medical record.
Groups:
- Exercise Group: Supervised, individualized exercise oncology program: Patients in the supervised exercise intervention group completed 12 weeks of prescribed, individualized exercise that aligned with American College of Sports Medicine (ACSM) exercise guidelines for cancer survivors. Total dose of exercise was once weekly, with cardiovascular, resistance training, and flexibility components. Cardiovascular exercise performed on a treadmill. The intensity level for the aerobic exercise began with 30 min at 30% of the individual's predicted VO2max, assessed by heart monitors. Each week, intensity progressed until the participant reached 45%. Strength training involved full body workout, with emphasis on all major muscle groups and employed machines, free weights, and tubing. Patients completed 3 sets of 10 repetitions for each exercise. Each exercise program was individualized for each patient, but included the following resistance exercises: chest press, seated row, overhead press, leg extension, leg curl, leg press. Resistance intensity was set at minimum of 30% of the individual's 1 Repetition Maximum1(RM), or when the patient felt sufficiently fatigued after 10 repetitions completed with proper form. As the patient's Rating of Perceived Exertion (RPE) values decreased with each exercise, intensity was progressively increased, accordingly. Flexibility training involved static stretching for 15-20 seconds at the completion of each workout. Each session lasted approximately 60 minutes.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Numbers of Breaks in Cancer Treatment
Description: Defined as missing 3 or more fractions due to patient condition, determined by electronic medical record
Time Frame: 12 weeks
Population: This data was not collected from the medical record. Study personnel could not determine from the medical record.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Cost of Emergency Room Visits
Description: Medical expenditure and utilization, for each time a patient utilized an emergency room visit for the purpose of managing health problems in addition to the planned cancer care, determined by electronic medical record.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Dollars ($)
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 129 | 122
Dollars ($) | 661 (210) | 989 (241)

4. Primary Outcome: Encounters
Description: Number of inpatient and outpatient hospital encounters, determined by electronic medical record
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: total number of encounters
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 129 | 122
total number of encounters | 7 (7) | 12 (6)

5. Primary Outcome: Cost of Total Unplanned Expenditures
Description: Number of hospital readmissions for the same presenting issue, determined by electronic medical record
Time Frame: 12 weeks
Population: "0" participants were analyzed because study personnel could not determine this from the electronic medical record.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Cost of Hospital Inpatient Care
Description: Hospital length of stay, in days, if applicable. Determined by electronic medical record.
Time Frame: 12 weeks
Population: "0" participants were analyzed because study personnel could not determine this from the EMR
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Cancer Treatment Adherence
Description: Percentage of patient adherence to their cancer treatment, determined by electronic medical record
Time Frame: 12 weeks
Population: This data was not collected from the medical record - "0" participants were analyzed because study personnel could not determine this from the medical record.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Cancer Treatment Symptom Management Medications
Description: Number of the different types of medications taken by patients for symptom management during their cancer treatment. Determined by electronic medical record.
Time Frame: 12 weeks
Population: as for outcome 7
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Cancer Treatment Related Side Effects
Description: Total number of cancer treatment related side effects
Time Frame: 12 weeks
Population: as for outcome 7
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Patient Rated Pain Score
Description: The Short Form-36 survey was used to measure pain. A high score defines a more favorable health state. Each item is scored on a 0 to 100 range, with the lowest and highest possible scores being 0 and 100, respectively.
Time Frame: 12 weeks, measured at the start of their exercise program during their initial assessment and at the 12-week follow-up re-assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 129 | 122
score on a scale
  At baseline | 50.4 (3.1) | 50.5 (3.16)
  At Follow-up (after 12 weeks of exercise training) | 62.3 (3.3) | 49.7 (3.2)

11. Primary Outcome: Cancer TreatmentTtolerance
Description: Measured by the Eastern Cooperative Oncology Group (ECOG) performance status score. Scale is from 0 to 5, with 0 being high functioning and no restriction and 5 being dead.
Time Frame: 12 weeks - ECOG performance status measurements were recorded at baseline and at the 12-week follow up appointment.
Population: Note that at baseline, there were 129 people in the control group (CG) and 122 people in the exercise group (EX). At follow up, there were 120 people in CG and 123 people in EX.
Measure: Number; unit: participants
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 129 | 122
participants
  Stage I Score 0-1 Baseline | 57 | 51
  Stage I Score 2 Baseline | 15 | 14
  Stage I Score 0-1 Follow-up: number analyzed (Participants) | 123 | 120
  Stage I Score 0-1 Follow-up | 46 | 45
  Stage I Score 2 Follow-up: number analyzed (Participants) | 123 | 120
  Stage I Score 2 Follow-up | 17 | 21
  Stage II Score 0-1 Baseline | 39 | 36
  Stage II Score 2 Baseline | 18 | 21
  Stage II Score 0-1 Follow-up: number analyzed (Participants) | 123 | 120
  Stage II Score 0-1 Follow-up | 36 | 21
  Stage II Score 2 Follow-up: number analyzed (Participants) | 123 | 120
  Stage II Score 2 Follow-up | 24 | 33

12. Primary Outcome: Quality of Life Measure: Utilizing McGill Quality of Life Survey and FACT-B Questionnaire
Description: McGill Quality of Life Survey:
  Physical Wellbeing (questions 1-4) - minimum score is 0, maximum score is 40. A higher score would be good and lower score would be bad.
  Social Wellbeing (questions 12, 14-16) - minimum score is 0, maximum score is 40. A higher score would be good and lower score would be bad.
  Emotional Wellbeing(questions 5-7, 13) - minimum score is 0 and maximum score is 40. A higher score would be bad and a lower score would be good Functional wellbeing (questions 8-11) - minimum score is 0, maximum score is 40. A higher score would be good and lower score would be bad.
  FACT-BREAST Survey:
  Minimum score is 0 and maximum is 148; 0 is not at all and 4 is very much, "good" or "bad" varies depending on the question; overall a higher score is good and a lower score is bad
Time Frame: Baseline was at the time of enrollment and follow up was after 12-weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 123 | 120
score on a scale
  Physical Well-Being at Baseline | 19.1 (1.7) | 19.2 (1.8)
  Physical Well-Being Post-Intervention | 23.1 (1.6) | 19.2 (1.9)
  Social Well-Being at Baseline | 19.6 (1.6) | 19.5 (1.7)
  Social Well-Being Post-Intervention | 23.1 (1.6) | 19.3 (1.6)
  Emotional Well-Being at Baseline | 18.7 (1.5) | 18.7 (1.4)
  Emotional Well-Being Post-Intervention | 20.2 (1.7) | 18.6 (1.2)
  Functional Well-Being at Baseline | 19.8 (1.5) | 19.9 (1.6)
  Functional Well-Being Post-Intervention | 23.2 (1.5) | 19.8 (1.7)
  FACT-Breast at Baseline | 98.2 (3.4) | 98.3 (3.5)
  FACT-Breast Post-Intervention | 114.2 (3.7) | 96.7 (3.5)

13. Secondary Outcome: Adherence Rate
Description: Exercise session adherence rate among the Exercise Group, collected from the Maple Tree Cancer Alliance participant records. Exercise session adherence rate was measured by dividing the total number of sessions scheduled by the total number of exercise sessions actually attended by the exercise group.
Time Frame: 12 weeks
Population: Because the control group did not participate in the exercise program, we did not calculate an adherence rate for this group.
Measure: Number; unit: percentage of session
Units Other Than Participants: exercise sessions
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 129 | 0
Number analyzed (exercise sessions) | 1548 | 0
percentage of session | 95 |

14. Secondary Outcome: Percentage of Participants Who Completed the Study (Attrition Rate)
Description: Exercise program attrition rate among the Exercise Group, collected from the Maple Tree Cancer Alliance participant records. Attrition was determined by calculating the percent of participants who completed the study by the total number of participants who started the study.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 129 | 122
percentage of participants | 95.3 | 98.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 12 weeks of the subjects' participation.
Arm/Group | Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/122
Other Adverse Events (participants affected / at risk) | 0/129 | 0/122

LIMITATIONS AND CAVEATS:
None to the study itself. Public funding and lack of resources have been identified as a significant barrier to national exercise oncology programs. Other known barriers include lack of general knowledge about the need to stay physically active during and after cancer therapy, qualified personnel, and available programs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT04106609/Prot_SAP_000.pdf